CLINICAL TRIAL: NCT04623567
Title: Efficacy Assessment of Chinese Herbal Medicine Jiangtang Tiaozhi Recipe Treating Participants With Glucose and Lipid Metabolism Disturbances and Associations Study Between Glucose and Lipid Metabolism Disturbances and Cardiovascular Risk Factors
Brief Title: Efficacy Assessment of Chinese Herbal Medicine Jiangtang Tiaozhi Recipe Treating Participants With Glucose and Lipid Metabolism Disturbances
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Jiaxing Tian, Attending Physician, Department of Endocrinology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD2020-4-4155
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Type2 Diabetes; Dyslipidemias
Keywords: type 2 diabetes mellitus; dyslipidemias; Jiangtang Tiaozhi Recipe; randomized controlled trial
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jiangtang Tiaozhi Recipe Group (Experimental): Jiangtang Tiaozhi formula granule (30g per bag), 1 bag per time, twice a day, take it with warm water after meals.
  Interventions: Drug: Jiangtang Tiaozhi recipe
- Metformin Group (Active Comparator): 500mg metformin tablet per time, 3 times a day, take it with meals.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Jiangtang Tiaozhi recipe — The Jiangtang Tiaozhi recipe is a combination of several Chinese herbs, which has been granted a patent (No. ZL 2013 1 0373659.7)
  Arms: Jiangtang Tiaozhi Recipe Group
Drug: Metformin — The metformin tablets (500mg) will be administrated.
  Other Names: Glucophage
  Arms: Metformin Group

SUMMARY:
This study is a randomized, positive drug parallel-controlled clinical trial in participants with glucose and lipid metabolism disturbances. A total of 96 participants will be recruited for the study, all of whom are diagnosed as type 2 diabetes mellitus combined with dyslipidemia. The subjects will be divided randomly into two groups and treated with either Jiangtang Tiaozhi Recipe or metformin. After 12 weeks of treatment, therapeutic effect of Jiangtang Tiaozhi Recipe will be evaluated based on the changes of HbA1c, fasting blood glucose, postprandial blood glucose, blood lipid, waist circumference, body mass index.

DETAILED DESCRIPTION:
The diagnosis criteria of type 2 diabetes mellitus are in accordance to 1999 World Health Organization (WHO) diabetes diagnostic criteria. The diagnosis criteria of dyslipidemia are based on the Guidelines for the Prevention and Treatment of Dyslipidemia in Chinese adults (2016, revision edition). The outcomes mainly include HbA1c, fasting blood glucose, postprandial blood glucose, body weight, waist circumference, blood lipid and TCM symptom score.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years at the time of their consent;
2. Diagnosed with type 2 diabetes;
3. TG≥1.7 mmol/L or LDL-C≥3.4 mmol/L;
4. BMI≥24.0 kg/m2 or male waist circumference≥90 cm, female waist circumference≥80 cm;
5. Failed to reach the normal standards of blood glucose and lipids after diet control and exercise therapy before enrollment;
6. TCM Syndrome differentiation as excess heat in the stomach and intestines syndrome;
7. Signed informed consent.

Exclusion Criteria:

1. Type 1 diabetes, gestational diabetes, other special types of diabetes.
2. Diabetic complications were the main symptoms, that is, patients with serious heart, lung, liver, kidney, brain complications or other serious primary diseases.
3. Patients with diabetic ketoacidosis, hyperosmolar nonketotic diabetic coma, severe infection, and surgery in recent one month.
4. Have a history of serious gastrointestinal diseases, or are suffering from serious gastrointestinal diseases, such as peptic ulcer, gastrointestinal bleeding, gastroparesis, pyloric stenosis, gastric shunt, etc..
5. Psychiatric patients, alcoholism and/or psychoactive substances, drug abusers and addicts.
6. Pregnant, preparing for pregnancy or lactation.
7. Patients who participated in other clinical studies within one month prior to participating in this study or were participating in other clinical studies.
8. According to the judgment of the researcher, other diseases or conditions that reduce the possibility of enrollment or complicate the enrollment, such as frequent changes in working environment and unstable living environment, are likely to cause loss of follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline HbA1c at 12 weeks | 0 week, 12 weeks
Changes from Baseline Fasting Blood Glucose at 4 weeks, 8 weeks,12 weeks | 0 week, 4 weeks, 8 weeks,12 weeks
Change from Baseline Postprandial Blood Glucose at 12 weeks | 0 week, 12 weeks
Change from Baseline Low Density Lipoprotein at 12 weeks | 0 week, 12 weeks
Change from Baseline Triglyceride at 12 weeks | 0 week, 12 weeks

SECONDARY OUTCOMES:
Changes from Baseline Body Mass Index at 4 weeks, 8 weeks,12 weeks | 0 week, 4 weeks, 8 weeks,12 weeks
Changes from Baseline Waist Circumference at 4 weeks, 8 weeks,12 weeks | 0 week, 4 weeks, 8 weeks,12 weeks
Change from Baseline Total Cholesterol at 12 weeks | 0 week, 12 weeks
Change from Baseline High Density Lipoprotein at 12 weeks | 0 week, 12 weeks
Change from Baseline TCM Symptom Score at 12 weeks | 0 week, 12 weeks

OTHER OUTCOMES:
Compositional and Functional Changes from Baseline Gut Microbiota at 12 weeks | 0 week, 12 weeks
Compositional and Functional Changes from Baseline Metabolites in blood and feces at 12 weeks | 0 week, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jiaxing Tian, PhD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu H, Fang X, Jin D, Miao R, Wei J, Zhao T, Dai D, Liao J, Wang J, Lian F, Tian J. Efficacy and Mechanism of the Jiangtang Tiaozhi Recipe in the Management of Type 2 Diabetes and Dyslipidaemia: A Clinical Trial Protocol. Front Pharmacol. 2022 Feb 4;13:827697. doi: 10.3389/fphar.2022.827697. eCollection 2022. PMID 35185579